CLINICAL TRIAL: NCT05389488
Title: A Randomized Pilot Study of the Efficacy of the OsciPulse System for the Reduction of Serum D-dimer
Brief Title: OsciPulse D-dimer Efficacy Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in funding
Sponsor: OsciFlex LLC (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSC-VTE-003
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Venous Thromboses; Ischemic Stroke
MeSH Terms: conditions — Venous Thrombosis; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control Arm (Active Comparator): Subjects will receive standard of care intermittent compression therapy using the current devices used in the clinical space.
  Interventions: Device: Flowtron ACS900
- Study Arm (Experimental): Subjects will receive compression therapy from the OsciPulse system.
  Interventions: Device: OsciPulse system

INTERVENTIONS:
Device: OsciPulse system — The OsciPulse system is a pneumatic compression system designed to provide intermittent compression to the limbs to augment venous blood flow.
  Arms: Study Arm
Device: Flowtron ACS900 — The Arjo Flowtron ACS900 intermittent pneumatic compression system provides compression the calf to augment venous blood flow.
  Arms: Control Arm

SUMMARY:
The purpose of this study is to assess the safety and efficacy of the OsciPulse System in reducing serum d-dimer levels in hospitalized ischemic stroke patients.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be screened for eligibility. Eligible and enrolled patients who have been admitted to the hospital for an ischemic stroke will be randomized in a non-blinded study to receive compression therapy from either standard-of-care intermittent compression garments, or the OsciPulse System. During the duration of the subject's hospital stay serum d-dimer levels will be monitored serially.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged ≥ 18 years old
2. Admitted to the Neuro Intensive Care Unit or Intermediate Neuro Care Unit with a diagnosis of ischemic stroke
3. Last known normal < 24 hours.
4. NIH stroke score ≥5
5. Weakness in at least one leg (≥ 1 point on the NIHSS lower extremity motor scores, items 6A and 6B)
6. Prescribed mechanical therapy for DVT prophylaxis.

Exclusion Criteria:

1. Inability or contraindication to applying IPC to both legs such as:

   * Evidence of bone fracture in lower extremities
   * Burns in the lower extremities, lacerations, ulcers, active skin infection or dermatitis,

     * ischemic limb in the legs at the site of IPC placement
   * Acute ischemia in the lower extremities
   * Severe peripheral vascular disease
   * Amputated foot or leg on one or two sides
   * Compartment syndrome
   * Severe lower extremity edema
   * Acute deep vein thrombosis
2. Subjects who received tPA therapy for their stroke
3. Pregnancy or within 6 weeks of postpartum period
4. Limitation of life support, life expectancy < 7 days, or in hospice care
5. A head-unit is unavailable for the first 24 hours or more
6. At the discretion of the attending physician and / or clinical team, the subject's participation in the study is believed not to be in the best interest of the subject.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Relative change in serum d-dimer levels | 7 days
  We will measure the change in serum d-dimer levels over time as a marker of venous coagulation.

SECONDARY OUTCOMES:
Device tolerability | 7 days
  We will measure the number of patients that are compliant with the treatment and quantify their experience with a questionnaire.

OTHER OUTCOMES:
Device Safety event rate | 7 days
  We will monitor for any device related adverse events - skin ulceration, DVT/PE, limb ischemia, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available following publication of the study results. The data will be available for 24 months.
Access Criteria: The data will be available to university or non-profit researchers.